CLINICAL TRIAL: NCT01339000
Title: A Multicenter Phase II Study of Enhancement of Immune Reconstitution and Vaccine Responses With Administration of Glyco-Recombinant Human IL-7(CYT107) in Older Subjects Following Chemotherapy
Brief Title: Improving the Immune System With Human IL-7 Vaccine in Older Subjects Who Have Had Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company supplying drug declared bankruptcy, thus there was no drug supply.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ronald Gress, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110146; 11-C-0146
Record Dates: First submitted 2011-04-19; First posted 2011-04-20 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer; Colon Cancer; Bladder Cancer
Keywords: Colorectal Cancer; Breast Cancer; Immunization; Immunocompromised Host; Bladder Cancer; Colon Cancer
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Urinary Bladder Neoplasms; Colorectal Neoplasms | interventions — Diphtheria-Tetanus Vaccine; Pneumococcal Vaccines; Hepatitis A Vaccines; Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A -Sequence 1 Immunizations (Experimental): Receive vaccine of Sequence 1 first, then vaccines of Sequence 2, 7 weeks later, after receiving interleukin-7 (IL-7)
  Interventions: Drug: Glycosylated Recombinant Human Interleukin-7; Biological: Diphtheria/Tetanus Vaccine; Biological: Polio Vaccine; Biological: Pneumococcal Vaccine; Biological: Hepatitis A Vaccine; Biological: Hepatitis B Vaccine
- Arm B - Sequence 2 Immunizations (Experimental): Receive vaccines of Sequence 2 first then vaccines of Sequence1, 7 weeks later, after receiving IL-7
  Interventions: Drug: Glycosylated Recombinant Human Interleukin-7; Biological: Diphtheria/Tetanus Vaccine; Biological: Polio Vaccine; Biological: Pneumococcal Vaccine; Biological: Hepatitis A Vaccine; Biological: Hepatitis B Vaccine

INTERVENTIONS:
Drug: Glycosylated Recombinant Human Interleukin-7 — Interleukin-7 (CYT 107) 20 microgram/kg / dose, by intramuscular (IM) injection
Biological: Diphtheria/Tetanus Vaccine — Diphtheria/Tetanus Vaccine will be administered according to the random schedule per protocol.
Biological: Polio Vaccine — Polio Vaccine will be administered according to the randomized schedule per protocol.
Biological: Pneumococcal Vaccine — Pneumococcal Vaccine will be administered according to the randomization schedule per protocol.
Biological: Hepatitis A Vaccine — Hepatitis A Vaccine will be administered according to the randomization schedule per protocol.
Biological: Hepatitis B Vaccine — Hepatitis B vaccine will be administered according to the randomization schedule per protocol.

SUMMARY:
Background: Drugs given to treat cancer (chemotherapy) can weaken the human immune system. But it can also become weaker because of aging. Interleukin (IL)-7, a molecule produced naturally in the body, can help improve the function of the immune system. Researchers want to study the effects of IL-7 on immune system function in two different groups of older people. One group will be people who have received vaccines before IL-7. The other group will be people who have received Vaccines after IL-7.

Objectives: To evaluate the effect of IL-7 on the immune system responses to vaccines in older people following chemotherapy.

Eligibility: People at least 60 years of age who have recently finished chemotherapy for breast, colon, or bladder cancer.

Design:

* People in the study will be screened with a physical examination, medical history, and blood tests. Other screening tests, such as tumor imaging, may also need to be performed.
* Everyone will receive a series of five different vaccines commonly used to prevent diseases. We will compare the responses of people in Sequence 1 who will receive vaccines before IL-7 with the responses of people in Sequence 2 who received the same vaccines after IL-7.
* The vaccines will be given randomly in two Arms at different times.

  * Arm 1: diphtheria and tetanus, polio, pneumonia (with two booster shots), hepatitis B (with two booster shots), and hepatitis A (with one booster shot),
  * Arm 2: hepatitis A (with one booster shot), hepatitis B (with two booster shots), pneumococcal (with two booster shots), diphtheria and tetanus, polio, pneumonia (with two booster shots)
* There are 5 vaccines to be given to each subject, following one of two randomly assigned sequences of vaccine administration (Sequence 1 or Sequence 2).
* The first vaccine arm contains the two diphtheria protein containing vaccines tetanus and diphtheria (Td) and pneumococcal conjugate 13 (PCV13) and polio. The second vaccine arm contains the Hepatitis A and Hepatitis B vaccines. Subjects will either get tetanus, diphtheria, polio, and pneumonia vaccines before IL-7 therapy (Sequence 1) or hepatitis A and hepatitis B vaccines before IL-7 therapy (Sequence 2). The response to vaccines will be evaluated 4 weeks after vaccination. This will be followed by IL-7 therapy, then administration of the other group of vaccines. Therefore, subjects on both arms will receive the same set of vaccines, just at different times with respect to IL-7 therapy.

DETAILED DESCRIPTION:
BACKGROUND:

* Interleukin-7 is a homeostatic cytokine with a critical role in lymphoid homeostasis through which it exerts its immune-restorative effects, particularly re-expansion of the naive and memory T cell subsets.
* The clinical implications of the kinetics, nature and extent of immune reconstitution defects following standard or ablative chemotherapy in older adults with cancer (in particular the lack of reconstitution of large pools naive T cell with broad repertoire diversity and of memory T cells) are not fully appreciated.
* As chemotherapy often induces only temporary complete or partial disease responses but no cure, candidates for novel immunotherapy strategies may be significantly impeded in their responses to active immunotherapy attempts, the therapeutic potential of which may be misjudged or altogether overlooked.
* Recombinant human interleukin-7 (rhIL-7) may play a role in immune reconstitution and immune enhancement in various circumstances of immune insufficiency in older individuals following chemotherapy or in the context of enhancing cancer immunotherapy or during immune senescence.

OBJECTIVES:

- Evaluate and quantify the impact of interleukin-7 (CYT107) therapy on specific immune responses to each vaccine (in particular to neo antigens) in older subjects following chemotherapy.

ELIGIBILITY:

* Adults over the age of 60.
* Diagnosis of non metastatic breast, bladder or colorectal cancer following adjuvant / neo-adjuvant chemotherapy.
* Completed a treatment with chemotherapy a minimum of 4 weeks prior to entry.
* Reasonable expectation that no chemotherapy will be given in the subsequent 6 months.

DESIGN:

* Subjects will be enrolled following the specific therapy for their respective diseases.
* Subjects will undergo immunizations with various antigens, randomized to be administered either before or after treatment with CYT107
* The vaccines, randomly assigned to be administered before CYT107 therapy are administered four weeks before the start of CYT107 therapy.
* CYT107 is administered once a week for 3 doses (20 microg/kg/dose) via intramuscular route (IM)
* The vaccines, randomly assigned to be administered after CYT107 therapy are administered 17 days after the first dose of CYT107 therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adults over the age of 60
* Documentation of positive diagnosis for any of the following:

  * Non metastatic breast carcinoma following neo-adjuvant chemotherapy and appropriate surgery or following adjuvant radio / chemotherapy.
  * Stage II or III colon carcinoma following appropriate surgery and adjuvant chemotherapy or following appropriate neoadjuvant chemoradiation/surgery and adjuvant chemotherapy.
  * Stage II bladder carcinoma following neo-adjuvant chemotherapy and appropriate surgery or following adjuvant chemotherapy. Patients with recurrent tumors are not eligible.
  * Appropriate therapy for each disease must be consistent with the latest National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines in Oncology available at the web site: http://www.nccn.org/professionals/physician_gls/f_guidelines.asp
  * Completed cancer specific therapy (including surgery, radiotherapy and/or chemotherapy) a minimum of 4 weeks prior to entry. (Subjects with hormone receptor positive breast carcinoma maintained on hormonal therapy following chemotherapy and radiation are eligible).
* Completed cancer specific therapy at most 6 months prior to entry.
* Reasonable expectation that no chemotherapy will be given in the subsequent 6 months (Principal Investigators (PIs) discretion).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times the upper limit of normal.
* Bilirubin < 1.5.
* Absolute Neutrophil Count greater than l000 / mm(3).
* Platelet count greater than 75K.
* International normalized ratio (INR)/partial thromboplastin time (PTT) within 1.5 times upper limit of normal (Common Terminology Criteria in Adverse Events (CTCAE) 4.0 grade 1 abnormality is acceptable)
* Serum creatinine within 1.5 times upper limit of normal (CTCAE 4.0 grade 1 abnormality is acceptable)
* Creatine phosphokinase (CPK) within 2.5 times upper limit of normal (CTCAE 4.0 grade 1 abnormality is acceptable)
* Serum albumin greater or equal to 3g/dl (CTCAE 4.0 grade 1 abnormality is acceptable)
* Serum electrolytes within normal limits (CTCAE 4.0 grade 1 abnormality is acceptable)
* Karnofsky performance status greater or equal to 70%.

EXCLUSION CRITERIA FOR ALL PARTICIPANTS:

* Significant heart disease defined as:

  * Significant coronary arterial disease
  * myocardial infarction in the last 6 months, angina in the previous 3 months,
  * Troponin elevation at level of myocardial infarction as defined by the manufacturer
  * Ischemic changes on electrocardiogram (ECG)
  * Atrio-ventricular block greater than 1st degree, in absence of pacemaker,
  * Corrected QT interval (QTc) greater than 480ms (CTCAE 4.0 grade 1 abnormality is acceptable),
  * History of ventricular arrhythmia,
  * Left Ventricular Ejection Fraction below the institutional limit of normal,
* Positive serology for human T-lymphotropic viruses, type 1 (HTLV I), human immunodeficiency virus (HIV), hepatitis A, hepatitis B, or hepatitis C infection including a positive hepatitis B serology indicative of previous immunization (i.e. hepatitis B surface antibody (HBs Ab) positive and hepatitis B core antibody (HBc Ab) negative)
* History of autoimmune disease: patients with vitiligo or endocrine disease controlled by replacement therapy including, diabetes, thyroid and adrenal disease may be enrolled
* Patients requiring chronic immunosuppressive therapy (including corticosteroids) for any medical condition,
* Splenomegaly or history of proliferative hematologic disease
* Prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation
* Inability or refusal to practice contraception during therapy (as physiologically relevant)
* History of medical or psychiatric disease which, in the view of the principal investigator, would preclude safe treatment
* Cognitive impairment
* Serious bleeding diathesis or those who are on therapeutic anticoagulation
* Previous exposure to Hepatitis A or B vaccines

Patients who received a tetanus and diphtheria (Td) or tetanus, diphtheria- acelluar, pertussis (Tdap) immunization in the previous 5 years,

* History of anaphylaxis or serious allergic reactions to previous administration of any of the vaccines
* Known hypersensitivity to any of the following: diphtheria toxoid, neomycin, polymixin B, streptomycin, 2 phenoxyethanol, formaldehyde, aluminum hydroxide, yeast
* Patients who had received one or more doses of the pneumococcal polysaccharide vaccine 23 (PPSV23) vaccine in the previous 12 months
* Inability to give informed consent

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Gress, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] BOWMAN BU Jr, PATNODE RA. NEUTRALIZATION OF BACTERIOPHAGE PHI-X174 BY SPECIFIC ANTISERUM. J Immunol. 1964 Apr;92:507-14. No abstract available. PMID 14139020
- [Background] Finkelstein MS, Uhr JW. Antibody formation. V. The avidity of gamma-M and gamma-G guinea pig antibodies to bacteriophage phi-x 174. J Immunol. 1966 Nov;97(5):565-76. No abstract available. PMID 5926449
- [Background] ROLFE U, SINSHEIMER RL. ANTIGENS OF BACTERIOPHAGE PHI-X174. J Immunol. 1965 Jan;94:18-21. No abstract available. PMID 14253517

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - Sequence 1 Immunizations: Receive vaccine of Sequence 1 first, then vaccines of Sequence 2, 7 weeks later, after receiving interleukin-7 (IL-7)
  Glycosylated Recombinant Human Interleukin-7: Interleukin-7 (CYT 107) 20 microgram/kg / dose, by intramuscular (IM) injection
  Diphtheria/Tetanus Vaccine: Diphtheria/Tetanus Vaccine will be administered according to the random schedule per protocol.
  Polio Vaccine: Polio Vaccine will be administered according to the randomized schedule per protocol.
  Pneumococcal Vaccine: Pneumococcal Vaccine will be administered according to the randomization schedule per protocol.
  Hepatitis A Vaccine: Hepatitis A Vaccine will be administered according to the randomization schedule per protocol.
  Hepatitis B Vaccine: Hepatitis B vaccine will be administered according to the randomization schedule per protocol.
Period: Overall Study
Arm/Group | Arm A - Sequence 1 Immunizations | Arm B - Sequence 2 Immunizations
Started | 1 (The patient received day 1, 29, 36, 43, 50, and 57 vaccines but did not receive interleukin-7 (IL-7)) | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — study closed due to lack of drug supply | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Sequence 1 Immunizations | Arm B - Sequence 2 Immunizations | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (0) |  | 61.3 (0)
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluate and Quantify the Impact of Interleukin-7 (CYT107) Therapy on Specific Immune Responses to Vaccines (in Particular to Neo Antigens) in Older Subjects Following Chemotherapy
Time Frame: 8 weeks
Population: Insufficient data was collected for any analysis to take place. The study was closed due to lack of drug supply.
Arm/Group | Arm A - Sequence 1 Immunizations | Arm B - Sequence 2 Immunizations
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Evaluate and Quantify the Impact of Interleukin-7 (CYT107) Therapy on the T Cell Receptor Diversity in Older Subjects Following Chemotherapy
Time Frame: 10 weeks
Population: Insufficient data was collected for any analysis to take place. The study was closed due to lack of drug supply.
Arm/Group | Arm A -Sequence 1 Immunizations | Arm B - Sequence 2 Immunizations
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Evaluate the Effects of Interleukin-7 (CYT107) Therapy on the Quality of T Cell Specific Responses by Multiparameter Flow Cytometry
Time Frame: 8 weeks
Population: Insufficient data was collected for any analysis to take place. The study was closed due to lack of drug supply.
Arm/Group | Arm A - Sequence 1 Immunizations | Arm B - Sequence 2 Immunizations
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Based on the First Two Primary Objectives, Consider and Discuss the Need for Larger Studies to Evaluate the Potential Benefit of Interleukin-7 (CYT107) Administration in a Broad, Mass Protection Strategy for an Aging Population
Time Frame: 1 year
Population: Insufficient data was collected for any analysis to take place. The study was closed due to lack of drug supply.
Groups:
- Arm A - Sequence 1 Immunizationa: Receive vaccine of Sequence 1 first, then vaccines of Sequence 2, 7 weeks later, after receiving interleukin-7 (IL-7)
  Glycosylated Recombinant Human Interleukin-7: Interleukin-7 (CYT 107) 20 microgram/kg / dose, by intramuscular (IM) injection
  Diphtheria/Tetanus Vaccine: Diphtheria/Tetanus Vaccine will be administered according to the random schedule per protocol.
  Polio Vaccine: Polio Vaccine will be administered according to the randomized schedule per protocol.
  Pneumococcal Vaccine: Pneumococcal Vaccine will be administered according to the randomization schedule per protocol.
  Hepatitis A Vaccine: Hepatitis A Vaccine will be administered according to the randomization schedule per protocol.
  Hepatitis B Vaccine: Hepatitis B vaccine will be administered according to the randomization schedule per protocol.
Arm/Group | Arm A - Sequence 1 Immunizationa | Arm B - Sequence 2 Immunizations
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 12 months
Measure: Number; unit: participants
Groups:
- Arm B - Sequence Immunizations: Receive vaccines of Sequence 2 first then vaccines of Sequence1, 7 weeks later, after receiving IL-7
  Glycosylated Recombinant Human Interleukin-7: Interleukin-7 (CYT 107) 20 microgram/kg / dose, by intramuscular (IM) injection
  Diphtheria/Tetanus Vaccine: Diphtheria/Tetanus Vaccine will be administered according to the random schedule per protocol.
  Polio Vaccine: Polio Vaccine will be administered according to the randomized schedule per protocol.
  Pneumococcal Vaccine: Pneumococcal Vaccine will be administered according to the randomization schedule per protocol.
  Hepatitis A Vaccine: Hepatitis A Vaccine will be administered according to the randomization schedule per protocol.
  Hepatitis B Vaccine: Hepatitis B vaccine will be administered according to the randomization schedule per protocol.
Arm/Group | Arm A - Sequence 1 Immunizations | Arm B - Sequence Immunizations
Number analyzed (Participants) | 1 | 0
participants | 0 |

ADVERSE EVENTS:
Arm/Group | Arm A - Sequence 1 Immunizations | Arm B - Sequence 2 Immunizations
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
The company supplying interleukin-7 (IL-7) declared bankruptcy, thus the study was closed due to lack of drug supply.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No